CLINICAL TRIAL: NCT04198961
Title: An Electronic Chart Intervention to Improve Safety for Patients on Chronic Opioid Therapy
Brief Title: Electronic Intervention to Chronic Opioid Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Huiqiong Deng, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-54148
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Opioid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic Intervention (Experimental): Individualized opioid taper and safety recommendations will be communicated to prescribers via an electronic medical record encrypted message.
  Interventions: Other: opioid prescribing

INTERVENTIONS:
Other: opioid prescribing — Individualized taper and safety recommendations will be communicated to prescribers via an electronic medical record encrypted message.

SUMMARY:
This pilot study will attempt to apply an electronic chart intervention to improve safety for patients on chronic opioid medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed long-term opioid therapy of doses greater than 90 morphine equivalent daily dose (MEDD)

Exclusion Criteria:

* Patients prescribed short-term opioid medications for acute pain (less than a 90-day supply over the past 120 days), sublingual buprenorphine, methadone maintenance for opioid use disorder or with oncology or palliative care diagnoses will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Change in the number of patients who receives naloxone prescription | baseline, 1, 3- and 6-months and 12 months
  Change in the number of patients who receives naloxone prescription
change of number of documentation about safety discussions | baseline, 1, 3- and 6-months and 12 months
  change of number of documentation about safety discussions
change of number of order for urine toxicology screening | baseline, 1, 3- and 6-months and 12 months
  change of number of order for urine toxicology screening
change of number of documentation of prescription drug monitoring program (CURES) results | baseline, 1, 3- and 6-months and 12 months
  change of number of documentation of prescription drug monitoring program (CURES) results
change of number of signed opioid informed consent forms | baseline, 1, 3- and 6-months and 12 months
  change of number of signed opioid informed consent forms

SECONDARY OUTCOMES:
Change in number of patients on long-term high risk doses of opioid pain medications | baseline, 1, 3- and 6-months and 12 months
  decreases in daily dose of opioids and number of patients on opioids ≥ 90mg MEDD

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiong Deng, MD, PHD, Principal Investigator — Stanford Univeristy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided